CLINICAL TRIAL: NCT05761431
Title: A Single-dose Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Octreotide Injection in Healthy Adult Subjects
Brief Title: A Single-dose Study of Octreotide Injection in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYHX2008-001
Record Dates: First submitted 2023-02-13; First posted 2023-03-09 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Injections; Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 5 mg cohort (Experimental): Subjects will be randomly assigned 4:1 to single dose of either SYHX2008（octreotide long-acting injection) or placebo at dose of 5 mg (8 active : 2 placebo).
  Interventions: Drug: SYHX2008 injection; Drug: Placebo to SYHX2008 injection
- 10 mg cohort (Experimental): Subjects will be randomly assigned 4:1 to single dose of either SYHX2008 or placebo at dose of 10 mg (8 active : 2 placebo).
  Interventions: Drug: SYHX2008 injection; Drug: Placebo to SYHX2008 injection
- 20 mg cohort (Experimental): Subjects will be randomly assigned 4:1 to single dose of either SYHX2008 or placebo at dose of 20 mg (8 active : 2 placebo).
  Interventions: Drug: SYHX2008 injection; Drug: Placebo to SYHX2008 injection
- 30 mg cohort (Experimental): Subjects will be randomly assigned 4:1 to single dose of either SYHX2008 or placebo at dose of 30 mg (8 active : 2 placebo).
  Interventions: Drug: SYHX2008 injection
- Octreotide long-acting release ( Sandostatin LAR®) 20 mg cohort (Experimental): Subjects will be treated with single dose of octreotide long-acting release ( Sandostatin LAR®) at dose of 20 mg.
  Interventions: Drug: Octreotide Acetate Microspheres for Injection injection
- Sandostatin® 0.1mg cohort (Experimental): Subjects will be treated with single dose of Sandostatin® at dose of 0.1mg.
  Interventions: Drug: Sandostatin ® injection

INTERVENTIONS:
Drug: SYHX2008 injection — Subcutaneous administration on Day 1.
  Arms: 10 mg cohort; 20 mg cohort; 30 mg cohort; 5 mg cohort
Drug: Octreotide Acetate Microspheres for Injection injection — Intramuscular administration on Day 1.
  Arms: Octreotide long-acting release ( Sandostatin LAR®) 20 mg cohort
Drug: Sandostatin ® injection — Subcutaneous administration on Day 1.
  Arms: Sandostatin® 0.1mg cohort
Drug: Placebo to SYHX2008 injection — Subcutaneous administration on Day 1.
  Arms: 10 mg cohort; 20 mg cohort; 5 mg cohort

SUMMARY:
This is a single-centre, single-dose, dose-escalation, placebo and positive drug-controlled Phase I clinical study in healthy Chinese subjects to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic profile of octreotide injection in healthy Chinese subjects.

DETAILED DESCRIPTION:
This single centre study will be comprised of 6 cohorts. The single ascending dose part is comprises of 4 cohorts（5 mg, 10 mg, 20 mg, 30 mg).

The other 2 cohorts are octreotide long-acting release ( Sandostatin LAR® ) 20 mg and Sandostatin® 0.1 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male and female subjects, 22-45 years of age, inclusive, at screening;
2. Body weight≥50 kg in male subjects or≥45 kg in female subjects, with BMI 19.0 - 28.0 kg/m^2 (inclusive);
3. Good health without history of cardiovascular vascular, liver, kidney, respiratory system, digestive, nervous, blood, immune, cancer, endocrine disease or any system diseases that have completely recovery or no clinical significance by investigator's assessment;
4. No clinically relevant findings in the physical examination, ECG, abdominal ultrasonography, vital signs, laboratory examination by investigator's assessment;
5. Informed consent documents signed by subjects prior the study, and subjects could be able to read, comprehend the procedure or the adverse reaction about the trial;
6. Subjects (including female and male subjects) have no pregnancy plan and sperm (egg) donation plan and voluntarily take effective contraceptive methods from signing the informed consent form until 3 months after administration of investigational product.

Exclusion Criteria:

1. The subject has a history of sensitivity (such as asthma, urticaria, eczema, etc), or has a known hypersensitivity to any of the test materials or related compounds, or has allergic constitution;
2. The female subject of childbearing potential, is pregnant (as based on test results in the screening period) or is breast feeding;
3. The subject with any one of HBsAg, hepatitis C antibody, anti-HIV antibody and antibody of treponema pallidum positive;
4. The subject with chronic or acute gastrointestinal disease (such as dyspepsia, gastro-oesophageal reflux, gastric bleeding or peptic ulcer, etc), or has a history of gallbladder disease (such as gallstone, cholecystectomy, etc) and other diseases;
5. The subject has a history of acupuncture syncope or blood phobia, or has difficulty with vein blood collection or venipuncture;
6. The subject has difficulty with subcutaneous administration;
7. The subject has a history of drug abuse or dependence, or has a positive result of drug abuse test in urine;
8. The subject intake more than 14 units alcohol within 3 months before administration of investigational product (1 unit=360 mL of beer, or 45 mL spirits, or 150 mL grape wine), or can't control to drink alcohol;
9. The subject smoke more than 5 cigarettes per day within 3 months before administration of investigational product, or smoke within 48h before administration of investigational product, or are unwilling to stop any tobacco products;
10. The subject has a history of hospitalization or surgical operation within 3 months before screening;
11. The subject has participated in other clinical trials within 3 months before administration of investigational product;
12. The subject donated blood or lost blood >400 mL (except female physiological period) within 3 months before screening;
13. The subject received prescription or non-prescription drugs within 28 days before administration of investigational product, including the drug effect on growth hormone and insulin-like growth factor (such as epinephrine, cholinergic drugs, etc); or received dietary supplements within 7 days before administration of investigational product (such as vitamin, protein powder, etc);
14. The subject with consumption of food or beverage containing caffeine or xanthine within 72 hours before administration of investigational product (such as coffee, tea, cola, chocolate, etc), or grapefruit fruit, or products containing grapefruit ingredients;
15. The subject has received any products containing alcohol within 48 hours before administration of investigational product or has a positive result of breath alcohol test;
16. According to the investigator's judgment, there are other situations that are not suitable for participating in this clinical trial.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Throughout the study period, with an average of 60 days.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 12 hour, 24 hour, 48 hour, 96 hour, 168 hour, 336 hour, 576 hour, 1008 hour, 1416 hour.
  AUC from pre-dose to time 't' (AUC[0-t]) and pre-dose to infinite time (AUC[0-infinity]) of Octreotide
Maximum plasma concentration (Cmax) | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 12 hour, 24 hour, 48 hour, 96 hour, 168 hour, 336 hour, 576 hour, 1008 hour, 1416 hour.
  Maximum octreotide plasma concentration (Cmax) of Octreotide
Time to maximum plasma concentration (Tmax) | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 12 hour, 24 hour, 48 hour, 96 hour, 168 hour, 336 hour, 576 hour, 1008 hour, 1416 hour.
  Time to maximum octreotide plasma concentration (Tmax) of Octreotide
Terminal elimination half-life (t1/2) | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 12 hour, 24 hour, 48 hour, 96 hour, 168 hour, 336 hour, 576 hour, 1008 hour, 1416 hour.
  Plasma decay half-life is the time measured for the octreotide plasma concentration to decrease by one half.
Apparent systemic clearance (CL/F) | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 12 hour, 24 hour, 48 hour, 96 hour, 168 hour, 336 hour, 576 hour, 1008 hour, 1416 hour.
  CL/F is the volume of plasma cleared of octreotide per unit time.
Apparent volume of distribution (Vz/F) | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 12 hour, 24 hour, 48 hour, 96 hour, 168 hour, 336 hour, 576 hour, 1008 hour, 1416 hour.
  Vz/F is the apparent volume of distribution of octreotide during the terminal elimination phase .
Insulin-like growth factor-1 (IGF-1) concentrations over time. | Pre-dose, 1 hour, 4 hour, 12 hour, 24 hour, 48 hour, 96 hour, 168 hour, 336 hour, 576 hour, 1008 hour, 1416 hour.
  IGF-1 levels will be collected over time to compare the suppressive ability of octreotide.

CONTACTS AND LOCATIONS:
Overall Officials: Yang NA Lin, PhD, Principal Investigator — Beijing Anzhen Hospital; Shan NA Jing, PhD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No